CLINICAL TRIAL: NCT04762290
Title: Dance for Children With Autism: a Therapeutic Intervention to Improve Motor Ability, Quality of Life, Social Communication, Perceived Physical Competence, and Self-efficacy
Brief Title: Dance for Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rujuta B. Wilson, MD, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20-001680-AM-00005
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Neurodevelopmental Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: The study model is a waitlist control. There is an active group and a waitlist control group.
Who Masked: Outcomes Assessor
Masking Description: Certain direct outcome measure assessors will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Group (Active Comparator): This group will receive the intervention in the first 10 weeks of the study. The intervention is a dance intervention that consists of a series of expressive movements.
  Interventions: Other: Dance
- Waitlist Control (Other): This group will receive the intervention in the second 10 weeks of the study (after the active group and after pre-post assessments in the first 10 weeks during the time of no intervention).
  Interventions: Other: Dance

INTERVENTIONS:
Other: Dance — The intervention is a series of expressive dance movements.
  Other Names: expressive movement

SUMMARY:
Motor impairments are prominent in individuals with autism spectrum disorder (ASD) and other neurodevelopment disorders, and these impairments often impact the individual's ability to engage in organized physical activity programs (OPA). While many studies have identified dance and creative movement to be retrospectively and anecdotally therapeutic, there remains a paucity of literature regarding outcomes associated with these programs, and specifically, their impact on (1) perceived and objective gross and fine motor skills, (2) perceived ability to succeed in related or divergent goals or tasks, (3) quality of life for affected individuals and their caregivers. (4) adaptive function and socialization, (5) social communication

This study explores the impact of organized dance and creative movement classes on children with autism (ages 8-12) and their caregivers. Participants will complete a set of surveys and assessments designed to measure the above metrics (labeled 1, 2, and 3) at their first study visit. This initial assessment is expected to take place within two weeks prior to beginning the intervention (either a wait period or a series of 1-hour dance classes, which children will attend weekly for 10 weeks). The second and final study visit will consist of a similar set of surveys and assessments designed to measure the same metrics within the two weeks following completion of the dance class series. Participants who have completed the wait period at this point will then begin their set of 10 weekly dance classes. Expected duration of participation in the study is no longer than 14 weeks in total.

DETAILED DESCRIPTION:
Motor impairments are prominent in individuals with autism spectrum disorder (ASD) and other neurodevelopment disorders, and these impairments often impact the individual's ability to engage in organized physical activity programs (OPA). While many studies have identified dance and creative movement to be retrospectively and anecdotally therapeutic, there remains a paucity of literature regarding outcomes associated with these programs, and specifically, their impact on (1) perceived and objective gross and fine motor skills, (2) perceived ability to succeed in related or divergent goals or tasks, (3) quality of life for affected individuals and their caregivers, (4) Adaptive function and socialization, (5) social communication.

This study explores the impact of organized dance and creative movement classes on children with autism (ages 8-12) and their caregivers. Participants will complete a set of surveys and assessments designed to measure the above metrics (labeled 1, 2,3, 4, 5) at their first study visit. This initial assessment is expected to take place within two weeks prior to beginning the intervention (either a wait period or a series of 1-hour dance classes, which children will attend weekly for 10 weeks). The second and final study visit will consist of a similar set of surveys and assessments designed to measure the same metrics within the two weeks following completion of the dance class series. Participants who have completed the wait period at this point will then begin their set of 10 weekly dance classes.

ELIGIBILITY:
Inclusion Criteria:

* There are no inclusion criteria based on gender, pregnancy/childbearing potential, race, ethnicity, or language spoken
* Children must be between the ages of 8 to 12
* A diagnosis of a autism
* Complex speech/fully verbal

Exclusion Criteria:

* Children younger than 8 years of age
* Children older than 12 years of age
* Children without a diagnosis of autism
* Children who are not fully verbal (i.e. phrased speech, single words, or non-speaking)
* Children who have previously participated in dance classes held by the Dance program called the Expressive Movement Initiative

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 35 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Movement Assessment Battery for Children Checklist | 10 minutes
  Motor questionnaire. Higher scores indicate a worse outcome
Vineland Adaptive Behavior Scale | 45 minutes
  A measure of adaptive behavior and motor skills. The minimum value is 21 and maximum value is 140. Higher scores indicate a better outcome.
Perceived Motor Competence Scale Parent Report | 5 minutes
  A measure of perceived motor skills in the child. Higher scores indicate a better outcome. Scores are based on a likert scale of 1-4. The minimum score is 18 and the maximum score is 72.
Perceived Motor Competence Scale Child Report | 5 minutes
  A measure of perceived motor skills in the child (participant). Higher scores indicate a better outcome. The minimum score is 13 and the maximum score is 52.
Brief Observation of Social Communication Change | 10 minutes
  A videotaped observational coding of a child's social communication behavior.
Parenting Stress Scale | 5 minutes
  Measure of factors related to caregiver stress
Lifespan Self-Esteem Scale | 2 minutes
  Measure of self-esteem/self-confidence
Autism Impact Measure | 10 minutes
  Measure of child's behaviors and the degree of impact on everyday functioning
Quantitative Gait Assessment | 10 minutes
  Direct motor measure in which the child walks across a mat with embedded sensors. The mat used in this study is the Zeno Walkway Gait Analysis System. This assessment includes self-regulated walking, fast walking, and standing balance.

SECONDARY OUTCOMES:
Social responsiveness scale | 15 minutes
  A measure of social communication and autism traits. Higher scores indicate a worse outcome. A total T-score of 76 or higher is considered severe and strongly associated with a clinical diagnosis of Autistic Disorder. T-scores of 66 through 75 are interpreted as indicating Moderate deficiencies in reciprocal social behavior that are clinically significant and lead to substantial interference in everyday social interactions. T-scores of 60 to 65 are in the Mild range and indicate mild to moderate deficits in social interaction.T scores of 59 and below are considered to be within typical limits and generally not associated with clinically significant ASD
Survey for adults | 10 minutes
  Measure of child's physical activity levels and engagement
Survey for children | 10 minutes
  measure of self physical activity levels and engagement

CONTACTS AND LOCATIONS:
Overall Officials: Rujuta B Wilson, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA David Geffen School of Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
At this time, there is not a plan to provide confidential individual participant data to other researchers. This study does not entail a medical condition or study of medication for a specific medical or genetic condition.

REFERENCES:
- [Derived] Anderson JT, Toolan C, Coker E, Singer H, Pham D, Jackson N, Lord C, Wilson RB. A novel dance intervention program for children and adolescents with developmental disabilities: a pilot randomized control trial. BMC Sports Sci Med Rehabil. 2024 May 14;16(1):109. doi: 10.1186/s13102-024-00897-3. PMID 38745176